CLINICAL TRIAL: NCT01552720
Title: Clinical Investigation of Chinese Patients With Aortic Dissection
Brief Title: Clinical Characteristics, Management and Outcomes of Chinese Patients With Acute Aortic Dissection
Acronym: CCMOCPAAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Yang Li, MD, MD, Xijing Hospital
Other Study IDs: XJHEART2012; CRAD201203 (Other Grant/Funding Number: 2011BAI11B00)
Record Dates: First submitted 2012-03-07; First posted 2012-03-13 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2012-03

CONDITIONS: Aortic Dissection
Keywords: aorta; dissection; feature
MeSH Terms: conditions — Aortic Dissection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Data reported by the international registry of acute aortic dissection (IRAD) in not sufficient to reflect clinical characteristics of acute aortic dissection in China. Moreover, clinical characteristics of Acute aortic dissection have not evaluated to data. The aim of this study is analyze changing trend of clinical characteristics of Chinese patients with acute aortic dissection.

DETAILED DESCRIPTION:
Acute aortic dissection is the most common aortic emergency, with an annual incidence of 3-5 cases per 100 000 population. About 50% of these patients are dead within 48 hours, if untreated. To assess the clinical manifestation, diagnosis, management, and outcomes of patients with AAD, the International Registry of Acute Aortic Dissection (IRAD) was established in 1996, and has grown to include about 2000 patients from 26 large referral centers to date. All patients from IRAD are caucasians from developed countries wiht advanced medical care, however, the proportion of Asian is very low. Data reported by the IRAD in not sufficient to reflect clinical characteristics of Acute aortic dissection in China. Clinical characteristics of Chinese patients with acute aortic dissection have not evaluated to data. The aim of this study is to analyze clinical characteristics of Chinese patients with acute aortic dissection and clinical trend of acute aortic dissection.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute aortic dissection
* Type A dissection
* Type B dissection
* Retrograde type B dissection

Exclusion Criteria:

* Aortic aneurysm
* Myocardial infarction
* Cerebral accident
* Active infection
* Unwillingness to cooperation with study procedures or follow-up visits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese patients suffering acute aortic dissection
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Dihua Yi, PhD, MD, Study Director — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- See also: database — http://www.epiedc.com